CLINICAL TRIAL: NCT03176979
Title: Emerging Tools in the Detection of Breast Cancer: Comparison of Contrast Enhanced Spectral Mammography With Digital Breast Tomosynthesis to Conventional Imaging Techniques Including Contrast Enhanced Magnetic Resonance Imaging and 2D Mammography With or Without Targeted Ultrasound
Brief Title: Contrast Enhanced Spectral Mammography With Digital Breast Tomosynthesis For Patients With Newly Diagnosed Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1B-16-3; NCI-2017-00778 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1B-16-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (CESM with DBT) (Experimental): Patients undergo a clinical breast examination and a diagnostic mammogram with or without targeted breast ultrasound to the index cancer as part of their standard of care preoperative work-up. As part of the research study, patients receive contrast agent IV and then undergo a CESM with DBT over 30 minutes. Patients also receive a contrast agent, gadolinium, IV and undergo bilateral breast CE-MRI over 10 minutes.
  Interventions: Other: Contrast Agent; Procedure: Digital Tomosynthesis Mammography; Procedure: Dual-Energy Contrast-Enhanced Digital Spectral Mammography

INTERVENTIONS:
Other: Contrast Agent — Given IV
  Other Names: Contrast; Contrast Drugs; contrast material; Contrast Medium
Procedure: Digital Tomosynthesis Mammography — Undergo CESM with DBT
  Other Names: DBT; Digital Breast Tomosynthesis; Digital Tomosynthesis of the Breast
Procedure: Dual-Energy Contrast-Enhanced Digital Spectral Mammography — Undergo CESM with DBT
  Other Names: Dual-Energy Contrast-Enhanced Digital Mammography (CEDM); Dual-Energy Contrast-Enhanced Digital Subtraction Mammography

SUMMARY:
This pilot clinical trial studies how well contrast enhanced spectral mammography works with digital breast tomosynthesis in imaging patients with newly diagnosed breast cancer. Contrast enhanced spectral mammography uses a special dye that is injected into the veins before mammogram images are taken. Digital breast tomosynthesis uses multiple x-ray pictures to produce a 3-dimensional rendering of the entire breast. Contrast enhanced spectral mammography with digital breast tomosynthesis may highlight areas of concern within the breast in more detail than a standard mammogram and improve the accuracy of tumor size.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the index lesion size (the largest diameter) from each of the four readings (standard of care 2 dimensional [D], magnetic resonance imaging [MRI], contrast enhanced spectral mammography [CESM], 3D) to gold standard index lesion size from surgical pathology (the largest diameter).

II. To document the additional ipsilateral and contralateral breast cancer lesions detected by the MRI, CESM, and 3D readings listed above.

OUTLINE:

Patients undergo a clinical breast examination and a diagnostic mammogram with or without targeted breast ultrasound to the index cancer as part of their standard of care preoperative work-up. As part of the research study, patients receive contrast agent intravenously (IV) and then undergo a CESM with digital breast tomosynthesis (DBT) over 30 minutes. Patients also receive a contrast agent, gadolinium, IV and undergo bilateral breast contrast enhanced (CE)-MRI over 10 minutes.

After completion of study, patients are followed up within 24-96 hours.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed breast cancer patients

Exclusion Criteria:

* Women with history of surgical, medical, or radiation therapy for breast cancer
* Women with renal failure or insufficiency
* Women with iodine contrast allergy
* Women with gadolinium contrast allergy
* Women who are pregnant, possibly pregnant, or lactating
* Women undergoing neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Index lesion size using the largest diameter | Baseline
  Intra-class correlation will be used to assess the agreement of index lesion size from each imaging reading to the gold standard (histopathology at surgery). Bland-Altman plot will be used to illustrate the pattern of difference between each reading and the gold standard.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Yamashita, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States